CLINICAL TRIAL: NCT02757300
Title: Incidence of Mucosal Injury Using Pharyngeal Packing in Surgery of the Nasal Sinuses
Brief Title: Mucosal Injury Using Pharyngeal Packing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study performer moved away
Sponsor: Marienhospital Osnabrück (Other)
Responsible Party: Principal Investigator, Saskia Jetten, P.D. Dr. med. M. Beiderlinden, Marienhospital Osnabrück
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mho 004
Record Dates: First submitted 2016-04-19; First posted 2016-05-02 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Sore Throat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypopharyngeal packing (Experimental): Patients with indication for surgery of the sinuses were randomly assigned to one of the two study groups.
  After standardized anaesthetic management and PONV prophylaxis routinely applied the patients were screened for mucosal injury on second postoperative day. Furthermore, the amount of analgetic and anti-emetic drugs and the severity of pain and PONV were recorded throughout the hospital stay.
  Interventions: Device: Hypopharyngeal packing
- Without hypopharyngeal packing (Active Comparator): Patients with indication for surgery of the sinuses were randomly assigned to one of the two study groups.
  After standardized anaesthetic management and PONV prophylaxis routinely applied the patients were screened for mucosal injury on second postoperative day. Furthermore, the amount of analgetic and anti-emetic drugs and the severity of pain and PONV were recorded throughout the hospital stay.
  Interventions: Device: Without Hypopharyngeal packing

INTERVENTIONS:
Device: Hypopharyngeal packing — After introduction and orotracheal intubation a hypopharyngeal packing soaked with Chlorhexidinbis (D-gluconat) is placed.
  Arms: Hypopharyngeal packing
Device: Without Hypopharyngeal packing — After introduction and orotracheal intubation the patient will pass the operation without hypopharyngeal packing with a short tip coming out the mouth to imitate a packing.
  Arms: Without hypopharyngeal packing

SUMMARY:
After approval of the Institutional Review Board and written patient´s informed consent patients with indication for surgery of the sinuses were randomly assigned to one of the two study groups. After standardized anaesthetic management and PONV prophylaxis routinely applied the patients were screened for mucosal injury on second postoperative day. Furthermore, the amount of analgetic and anti-emetic drugs and the severity of pain and PONV were recorded throughout the hospital stay.

DETAILED DESCRIPTION:
Aim of the study

Post-operative nausea and vomiting (PONV) is a complication of anaesthesia and responsible for malaise of surgical patients. Furthermore, PONV has been shown causing additive costs due to anti-emetic drugs and prolonged hospitalisation. The occurrence of PONV is multifactorial. Beside individual patients factors, opioid use and type of surgery seem to be responsible for occurrence of PONV. Especially, sinus surgery carries a high risk of PONV. Blood from the operation site entering the stomach has been discussed the potential cause for PONV in this specific patient population.

Therefore, hypopharyngeal packing following orotracheal intubation is a common clinical practice to prevent blood passing through the esophagus and so to lower the incidence of PONV.

Unfortunately, there are limited data data supporting the effectiveness of this procedure. In contrast, some references suggest that hypopharyngeal packing may be associated with postoperative mucosal injury and sore throat with high impact on patients´ well-being.

To evaluate the usefulness and safety of hypopharyngeal packing the investigators perform prospective randomized study with the following objective:

1. Does pharyngeal packing during sinus surgery increase the incidence of mucosal injury?

ELIGIBILITY:
Inclusion Criteria:

* Surgery of the sinuses
* Patients over 18 years of age
* Duration of surgery > 1h

Exclusion Criteria:

* Refusal of the patient
* Patients under 18 years of age
* Chemotherapy with antiemetic medication
* Combined surgery (for example tonsillectomie and sinus surgery)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of mucosal injury | Second postoperative day
  Incidence and severity of mucosal injury evaluated by NRS-Scores and a colleague of the ENT department blinded to intra-operative management

CONTACTS AND LOCATIONS:
Overall Officials: Martin Beiderlinden, PD, Study Director — Marienhospital Osnabrück

IPD SHARING:
Plan to Share IPD: Undecided